CLINICAL TRIAL: NCT00992264
Title: Optimizing an Online Motivational Tobacco Cessation Program
Brief Title: 'Questions About Quitting' Smoking Cessation Trial
Acronym: Q2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01CA138598 (NIH)
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Smoking
Keywords: Cigarette Smoking; Health Behavior; Intervention Studies; Personal Communication
MeSH Terms: conditions — Smoking; Cigarette Smoking; Health Behavior; Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Message Tone (Experimental): Prescriptive or Motivational
  Persons are randomized to receive intervention content written in either a prescriptive or motivational tone.
  Interventions: Behavioral: Message Tone
- Testimonials (Experimental): Persons are randomized to receive a personally tailored testimonial or not.
  Interventions: Behavioral: Testimonials
- Navigation (Experimental): Dictated or Non-Dictated
  Persons are randomly assigned to be able to freely navigate the website or to have their navigation of the website pre-determined based on their baseline readiness to quit smoking.
  Interventions: Behavioral: Navigation
- Proactive Outreach (Experimental): Email or No-Email communication
  Persons are randomized to receive periodic email reminders to return to the intervention website or not.
  Interventions: Behavioral: Proactive Outreach

INTERVENTIONS:
Behavioral: Message Tone — All participants receive an tailored, online smoking cessation program. Participants in this intervention group either receive content written in a prescriptive tone or a motivational tone.
  Arms: Message Tone
Behavioral: Navigation — Persons in this arm either have their ability to navigate the site dictated for them based on their readiness to quit smoking or they are able to freely navigate through the website.
  Arms: Navigation
Behavioral: Proactive Outreach — Persons receive periodic, proactively delivered email reminders to visit the intervention website.
  Arms: Proactive Outreach
Behavioral: Testimonials — People receive a personally-tailored testimonial as part of their online smoking cessation program.
  Arms: Testimonials

SUMMARY:
The current study tested the effectiveness of four potentially important tailoring factors (decisional framework, self-efficacy, navigation autonomy, and proactive outreach) in the context of an online motivational intervention for smoking cessation. A fifth factor was originally planned by dropped during intervention development due to confounds with the other planned factors. Information learned from this study will inform how to best design an online interventions for smoking cessation. Participants were recruited from a large, regional U.S. health plan. Using a full factorial design to screen for important main effects and 2-way interactions, participants were randomized to receive one of 16 different experimental factor combinations and followed for one year to assess program impact on smokers' use of empirically-validated cessation treatment and abstinence.

DETAILED DESCRIPTION:
The current study is a factorial screening experiment, consistent with the Multiphase Optimization Strategy. Participants were randomly assigned to one of 16 different combinations of the 4 experimental factors. Each factor was explored on 2 contrasting levels. Each contrasting factor level was then compared to the other, resulting in 4 analytic arms. Within each arm, all participants (n = 1865) were analyzed to determine the relative effect of each contrasting factor level on the primary and secondary outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

* Member of Group Health Cooperative
* Currently Smoking at Least 5 Cigarettes/Day
* Access to Email and the Internet
* Read and Write English
* 18 years or older
* Not currently receiving tobacco cessation treatment
* Capable of participating in online and phone surveys

Exclusion Criteria:

* Persons will be excluded if they do not meet above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1865 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer B McClure, PhD, Principal Investigator — Group Health Research Institute
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Background] McClure JB, Derry H, Riggs KR, Westbrook EW, St John J, Shortreed SM, Bogart A, An LC. Questions about quitting (Q2): design and methods of a Multiphase Optimization Strategy (MOST) randomized screening experiment for an online, motivational smoking cessation intervention. Contemp Clin Trials. 2012 Sep;33(5):1094-102. doi: 10.1016/j.cct.2012.06.009. Epub 2012 Jul 4. PMID 22771577
- [Result] McClure JB, Shortreed SM, Bogart A, Derry H, Riggs K, St John J, Nair V, An L. The effect of program design on engagement with an internet-based smoking intervention: randomized factorial trial. J Med Internet Res. 2013 Mar 25;15(3):e69. doi: 10.2196/jmir.2508. PMID 23529377
- [Result] McClure JB, Peterson D, Derry H, Riggs K, Saint-Johnson J, Nair V, An L, Shortreed SM. Exploring the "active ingredients" of an online smoking intervention: a randomized factorial trial. Nicotine Tob Res. 2014 Aug;16(8):1129-39. doi: 10.1093/ntr/ntu057. Epub 2014 Apr 11. PMID 24727369
- [Derived] Shortreed SM, Bogart A, McClure JB. Using multiple imputations to accommodate time-outs in online interventions. J Med Internet Res. 2013 Nov 21;15(11):e252. doi: 10.2196/jmir.2781. PMID 24263289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Group Health, a large, non-profit health plan in the US Pacific Northwest. Data were collected between May 2010 and November 2012. All intervention and data collection occurred online.
Groups:
- Randomization Arm 1: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [prescriptive], navigation [dictated], proactive emails [yes], and testimonials [yes]
- Randomization Arm 2: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [prescriptive], navigation [not dictated], proactive emails [yes], and testimonials [yes]
- Randomization Arm 3: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [prescriptive], navigation [dictated], proactive emails [no], and testimonials [yes]
- Randomization Arm 4: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [prescriptive], navigation [not dictated], proactive emails [no], and testimonials [yes]
- Randomization Arm 5: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [prescriptive], navigation [dictated], proactive emails [yes], and testimonials [no]
- Randomization Arm 6: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [prescriptive], navigation [not dictated], proactive emails [yes], and testimonials [no]
- Randomization Arm 7: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [prescriptive], navigation [dictated], proactive emails [no], and testimonials [no]
- Randomization Arm 8: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [prescriptive], navigation [not dictated], proactive emails [no], and testimonials [no]
- Randomization Arm 9: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [motivational], navigation [dictated], proactive emails [yes], and testimonials [yes]
- Randomization Arm 10: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [motivational], navigation [not dictated], proactive emails [yes], and testimonials [yes]
- Randomization Arm 11: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [motivational], navigation [dictated], proactive emails [no], and testimonials [yes]
- Randomization Arm 12: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [motivational], navigation [not dictated], proactive emails [no], and testimonials [yes]
- Randomization Arm 13: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [motivational], navigation [dictated], proactive emails [yes], and testimonials [no]
- Randomization Arm 14: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [motivational], navigation [not dictated], proactive emails [yes], and testimonials [no]
- Randomization Arm 15: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [motivational], navigation [dictated], proactive emails [no], and testimonials [no]
- Randomization Arm 16: Persons in this group are randomized to the following combination of each of the experimental factors: message tone [motivational], navigation [not dictated], proactive emails [no], and testimonials [no]
Period: Overall Study
Arm/Group | Randomization Arm 1 | Randomization Arm 2 | Randomization Arm 3 | Randomization Arm 4 | Randomization Arm 5 | Randomization Arm 6 | Randomization Arm 7 | Randomization Arm 8 | Randomization Arm 9 | Randomization Arm 10 | Randomization Arm 11 | Randomization Arm 12 | Randomization Arm 13 | Randomization Arm 14 | Randomization Arm 15 | Randomization Arm 16
Started | 116 | 116 | 117 | 117 | 117 | 117 | 116 | 117 | 116 | 116 | 117 | 117 | 116 | 117 | 117 | 116
Completed | 116 (All enrolled participants were included in the final intent to treat analytic sample.) | 116 (All enrolled participants were included in the final intent to treat analytic sample.) | 117 (All enrolled participants were included in the final intent to treat analytic sample.) | 117 (All enrolled participants were included in the final intent to treat analytic sample.) | 117 (All enrolled participants were included in the final intent to treat analytic sample.) | 117 (All enrolled participants were included in the final intent to treat analytic sample.) | 116 (All enrolled participants were included in the final intent to treat analytic sample.) | 117 (All enrolled participants were included in the final intent to treat analytic sample.) | 116 (All enrolled participants were included in the final intent to treat analytic sample.) | 116 (All enrolled participants were included in the final intent to treat analytic sample.) | 117 (All enrolled participants were included in the final intent to treat analytic sample.) | 117 (All enrolled participants were included in the final intent to treat analytic sample.) | 116 (All enrolled participants were included in the final intent to treat analytic sample.) | 117 (All enrolled participants were included in the final intent to treat analytic sample.) | 117 (All enrolled participants were included in the final intent to treat analytic sample.) | 116 (All enrolled participants were included in the final intent to treat analytic sample.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1865 participants were enrolled and randomized. For the analyses, participants assigned to each contrasting level of each of the 4 experimental factors were compared against one another. Thus, 1865 people were in each analytic arm in this factorial screening experiment.
Groups:
- Randomization Arm: 1: Persons assigned to this arm received the following intervention combination: Tone [prescriptive], Navigation [dictated], proactive emails [yes], and testimonials [yes].
- Radndomization Arm: 2: Persons assigned to this arm received the following intervention combination: Tone [prescriptive], Navigation [not dictated], proactive emails [yes], and testimonials [yes].
- Randomization Arm: 3: Persons assigned to this arm received the following intervention combination: Tone [prescriptive], Navigation [dictated], proactive emails [no], and testimonials [yes].
- Randomization Arm: 4: Persons assigned to this arm received the following intervention combination: Tone [prescriptive], Navigation [not dictated], proactive emails [no], and testimonials [yes].
- Randomization Arm: 5: Persons assigned to this arm received the following intervention combination: Tone [prescriptive], Navigation [dictated], proactive emails [yes], and testimonials [no].
- Randomization Arm: 6: Persons assigned to this arm received the following intervention combination: Tone [prescriptive], Navigation [not dictated], proactive emails [yes], and testimonials [no].
- Randomization Arm: 7: Persons assigned to this arm received the following intervention combination: Tone [prescriptive], Navigation [dictated], proactive emails [no], and testimonials [no].
- Randomization Arm: 8: Persons assigned to this arm received the following intervention combination: Tone [prescriptive], Navigation [not dictated], proactive emails [no], and testimonials [no].
- Randomization Arm: 9: Persons assigned to this arm received the following intervention combination: Tone [motivational], Navigation [dictated], proactive emails [yes], and testimonials [yes].
- Randomization Arm: 10: Persons assigned to this arm received the following intervention combination: Tone [motivational], Navigation [not dictated], proactive emails [yes], and testimonials [yes].
- Randomization Arm: 11: Persons assigned to this arm received the following intervention combination: Tone [motivational], Navigation [dictated], proactive emails [no], and testimonials [yes].
- Randomization Arm: 12: Persons assigned to this arm received the following intervention combination: Tone [motivational], Navigation [not dictated], proactive emails [no], and testimonials [yes].
- Randomization Arm: 13: Persons assigned to this arm received the following intervention combination: Tone [motivational], Navigation [dictated], proactive emails [yes], and testimonials [no].
- Randomization Arm: 14: Persons assigned to this arm received the following intervention combination: Tone [motivational], Navigation [not dictated], proactive emails [yes], and testimonials [no].
- Randomization Arm: 15: Persons assigned to this arm received the following intervention combination: Tone [motivational], Navigation [dictated], proactive emails [no], and testimonials [no].
- Randomization Arm: 16: Persons assigned to this arm received the following intervention combination: Tone [motivational], Navigation [not dictated], proactive emails [no], and testimonials [no].
- Total: Total of all reporting groups
Arm/Group | Randomization Arm: 1 | Radndomization Arm: 2 | Randomization Arm: 3 | Randomization Arm: 4 | Randomization Arm: 5 | Randomization Arm: 6 | Randomization Arm: 7 | Randomization Arm: 8 | Randomization Arm: 9 | Randomization Arm: 10 | Randomization Arm: 11 | Randomization Arm: 12 | Randomization Arm: 13 | Randomization Arm: 14 | Randomization Arm: 15 | Randomization Arm: 16 | Total
Number analyzed (Participants) | 116 | 116 | 117 | 117 | 117 | 117 | 116 | 117 | 116 | 116 | 117 | 117 | 116 | 117 | 117 | 116 | 1865
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 111 | 108 | 110 | 111 | 110 | 111 | 108 | 108 | 108 | 112 | 109 | 111 | 114 | 113 | 110 | 109 | 1763
  >=65 years | 5 | 8 | 7 | 6 | 7 | 6 | 8 | 9 | 8 | 4 | 8 | 6 | 2 | 4 | 7 | 7 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.34 (14.50) | 44.06 (14.95) | 42.83 (15.06) | 45.93 (13.82) | 43.49 (14.34) | 43.84 (14.39) | 45.19 (14.6) | 44.33 (15.05) | 44.56 (15.43) | 43.82 (14.24) | 46.09 (14.75) | 45.03 (14.26) | 42.29 (15.07) | 43.69 (14.95) | 44.39 (14.95) | 43.99 (14.97) | 44.2 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 79 | 76 | 66 | 39 | 76 | 73 | 69 | 74 | 77 | 72 | 76 | 65 | 69 | 76 | 77 | 1139
  Male | 41 | 37 | 41 | 51 | 78 | 41 | 43 | 48 | 42 | 39 | 45 | 41 | 51 | 48 | 41 | 39 | 726
Region of Enrollment [Number; unit: participants]
  United States | 116 | 116 | 117 | 117 | 117 | 117 | 116 | 117 | 116 | 116 | 117 | 117 | 116 | 117 | 117 | 116 | 1865

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: 7 day point prevalent abstinence
Time Frame: 12 months
Population: Missing data imputed, so all enrolled participants were included in the final intent to treat analytic sample.
Measure: Number; unit: percentage of abstinent participants
Groups:
- Message Tone: Prescriptive: Persons in the 'active' comparison group received website content written in a prescriptive message tone.
  Persons in the comparison group received content written in a motivational message tone.
- Testimonials: Persons in the 'active' comparison group were randomized to receive a personally tailored testimonial.
  Persons in the comparison group did not receive the testimonial content.
- Navigation: Dictated: Persons in the 'active' comparison group had their navigation through the website dictated based on their baseline readiness to quit smoking.
  Persons in the comparison group could freely navigate the website.
- Proactive Outreach: Persons in the active comparison group were randomized to receive periodic email reminders to return to the intervention website.
  Persons in the comparison group did not receive proactive email reminders.
Arm/Group | Message Tone: Prescriptive | Testimonials | Navigation: Dictated | Proactive Outreach
Number analyzed (Participants) | 1865 | 1865 | 1865 | 1865
percentage of abstinent participants
  Smoking prevalence: 'active' intervention grp | 13.0 | 13.8 | 14.5 | 13.3
  smoking prevalence: comparison group | 14.5 | 13.6 | 13.0 | 14.2
Statistical Analysis 1: Comparison: Message Tone: Prescriptive; Comparison of persons assigned to Prescriptive message tone (n = 932) against persons assigned to Motivational message tone (n = 933); Test type: Superiority or Other; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.51 to 1.51] — OR for smoking abstinence at 12 months in intent to treat sample. Participants receiving content written in a Prescriptive tone were compared against persons receiving content in a Motivational tone (ref group)
Statistical Analysis 2: Comparison: Testimonials; Comparison of persons assigned to Testimonials (n = 933) against persons assigned to receive no testimonials (n = 932); Test type: Superiority or Other; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.66 to 1.91] — OR for smoking abstinence at 12 months when persons who randomly received a Testimonial were compared against persons receiving No Testimonial (ref group)
Statistical Analysis 3: Comparison: Navigation: Dictated; Comparison of persons assigned to the Dictated Navigation arm (n = 934) against persons assigned to assigned free navigation of the website (n = 931); Test type: Superiority or Other; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.70 to 2.02] — OR for smoking abstinence at 12 months when persons assigned to Dictated navigation were compared to those not assigned to Dictated navigation (ref group)
Statistical Analysis 4: Comparison: Proactive Outreach; Comparison of persons assigned to Proactive Email Outreach (n = 933) against persons assigned to receive No Proactive Email Outreach (n = 932); Test type: Superiority or Other; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.43 to 1.30] — OR for smoking abstinence at 12 months when persons assigned to receive Proactive Email reminders were compared against persons who received No Emails (ref group)

2. Primary Outcome: Treatment Utilization for Smoking Cessation
Description: confirmed use of pharmacotherapy or enrollment in health plan-sponsored counseling program
Time Frame: 12 months
Population: Twenty-seven participants were excluded for not being enrolled in the health plan during the study period and not having access to the provided adjunct treatment.
Measure: Number; unit: % of participants using adjunct treatmen
Groups:
- Proactive Emails: Persons in the active comparison group were randomized to receive periodic email reminders to return to the intervention website.
  Persons in the comparison group did not receive proactive email reminders.
Arm/Group | Message Tone: Prescriptive | Testimonials | Navigation: Dictated | Proactive Emails
Number analyzed (Participants) | 1838 | 1838 | 1838 | 1838
% of participants using adjunct treatmen
  Treatment utilization: % in active intervention | 26.1 | 25.3 | 26.0 | 23.7
  treatment utilization: % in comparison group | 25.8 | 26.6 | 25.9 | 28.2
Statistical Analysis 1: Comparison: Message Tone: Prescriptive vs Testimonials; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Odds Ratio, log = 0.94, 95% CI 2-sided [0.62 to 1.43] — OR for use of adjunct treatment at 12 months when persons assigned to Prescriptive Tone were compared to persons assigned to receive content in a Motivational Tone (ref group)
Statistical Analysis 2: Comparison: Testimonials; Comparison of persons assigned to Testimonials (n = 933) against persons assigned to receive no testimonials (n = 932); Test type: Superiority or Other; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.46 to 1.07] — OR for use of adjunct treatment at 12 months when persons assigned to receive a Testimonial were compared to persons assigned to receive No Testimonial (ref group)
Statistical Analysis 3: Comparison: Navigation: Dictated; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.51 to 1.18] — OR for use of adjunct treatment at 12 months when persons assigned to Dictated Navigation were compared to persons not assigned to Dictated Navigation (ref group)
Statistical Analysis 4: Comparison: Proactive Emails; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.44 to 1.03] — OR for use of adjunct treatment at 12 months when persons assigned to Proactive Email reminders were compared to persons not assigned to receive Proactive Email reminders (ref group)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from May 2010 until November 2012, the time during which participants were actively enrolled in this trial.
Description: Participants were instructed to contact study staff in the event of adverse events, including changes in their health or medical status. Other potential adverse events (e.g., breach of confidentiality) were monitored by study staff.
Groups:
- Testimonials: Testimonial or No Testimonial
  Persons are randomized to receive a personally tailored testimonial or not.
Arm/Group | Message Tone | Testimonials | Navigation | Proactive Outreach
Serious Adverse Events (participants affected / at risk) | 0/1865 | 0/1865 | 0/1865 | 0/1865
Other Adverse Events (participants affected / at risk) | 0/1865 | 0/1865 | 0/1865 | 0/1865

LIMITATIONS AND CAVEATS:
The study was powered to detect differences between each factor level of 5% or more.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No